CLINICAL TRIAL: NCT06615427
Title: Delivered and Assessed FiO2 in Neonates With Respiratory Distress and Treated With Bubble-CPAP at a Neonatal Intensive Care Unit in Hanoi, Vietnam
Brief Title: FiO2 Delivered With Neonatal bCPAP
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Göteborg University (Other); Hanoi Medical University (Other); Hanoi Obstetrics and Gynecology Hospital (Other)
Responsible Party: Principal Investigator, Thomas Drevhammar, Ass. prof. (Docent), Karolinska Institutet
Other Study IDs: 2024-05506-01
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2024-09

CONDITIONS: Respiratory Distress Syndrome (RDS); Infant, Premature, Diseases; Infant, Newborn, Diseases
Keywords: Continuous Positive Airway Pressure; Respiratory Therapy
MeSH Terms: conditions — Respiratory Distress Syndrome; Infant, Premature, Diseases; Infant, Newborn, Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infant treated with bubble CPAP and receiving blended air/oxygen

SUMMARY:
Continuous positive airway pressure (CPAP) is the mainstay of treatment recommended for preterm infants with respiratory distress syndrome in all resource contexts. Many of the available bubble CPAP machines in low- and middle-income contexts mix flows of air and oxygen. These are adjusted by two separate rotameters (flowmeters) and estimate FiO2 delivery. Medical decisions regarding interventions to sick neonates such as need for intubation or surfactant administration are in large part dependant on a reliable estimation of FiO2-delivery. The aim of this study is to evaluate the accuracy of FiO2 delivered by bubble-CPAP machines with separate oxygen and air rotameters in patients at a neonatal intensive care unit (NICU) in Hanoi.

DETAILED DESCRIPTION:
This is a cross-sectional observational study. The patient population will be a convenience sample with patients recruited when investigators are available, and the measurement is possible without interrupting planned care. There is no intervention apart from measurements of FiO2 in the breathing circuit and parents will be given the opportunity to decline participation. The study aims to include FiO2 measurements from bCPAP machines in use where the infants have stable spontaneous breathing and not expected to need urgent interventions. The main outcomes of the study are FiO2 displayed by the analyzer (chemical sensor), FiO2 recorded compared to FiO2 assessed from the rotameter flow using the conversion table. The clinicians estimating the rotameter flows are blinded to the delivered FiO2.

There are 22 bubble CPAP machines in the NICU. We aim to collect four or five measurements on each machine at a range of FiO2-levels generating a total of approximately 100 measurements. Differences in FiO2 of 0.04 would be considered clinically relevant, since it might have implication for decision of surfactant treatment or intubation. FiO2 accuracy will be investigated by comparing paired samples from visual assessed FiO2 and measured FiO2 (electrochemical sensor) by appropriate statistical tests. Variation between and within the two types of CPAP machines will be described. Analysis will also describe accuracy at different FiO2 levels and variance of accuracy between clinicians' bedside estimates.

The main application for ethical approval of the study will be to the Ethical Review Board at Phu San Hanoi Hospital. Analysis and data will be handled by researchers affiliated with Karolinska Institutet, and a second application will be filed at the Swedish Ethical Review Authority.

The risk for an infant participating in the study is minimal. Only infants with stable breathing will be included and measuring an infant is short with two brief interruptions in CPAP treatment. Pauses and interruptions of CPAP is common during normal care, for example when the nasal interfaces are repositioned, nares cleaned or tubes replaced. The infant is not moved and there is no handling of the infant or tests performed. Routine monitoring will be in place. The study takes place in the neonatal intensive care ward where there is immediate access to equipment and staff experienced with life support if an infant is sick. In that case the measurement can be immediately stopped without problems for the infant or the study.

For an infant there are no advantages or disadvantages with participating in the study. If the measured FiO2 deviates and this will affect management, the staff will be notified. This could for example be decisions regarding surfactant or mechanical ventilation. This is a potential advantage for the individual patients.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Phu San Hanoi Hospital Neonatology Unit
* Bubble CPAP support with added O2
* ≥28 weeks GA
* Stable spontaneous breathing
* Investigation team available

Exclusion Criteria:

* Unstable infants in need of urgent intervention
* Major congenital malformation
* Known syndrome or neuromuscular disorder
* Circulatory instability with inotropes
* Recently extubated (<24 h)
* Recent large surgical procedure (<5 days)

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study aims to include FiO2 measurements from bCPAP machines in use where the infants have stable spontaneous breathing and not expected to need urgent interventions.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-09-28 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
FiO2 delivered | 5 minutes
  FiO2 in breathing circuit using an oxygen sensor
FiO2 estimated | 5 minutes
  FiO2 in breathing circuit estimated from flow meters by clinician

OTHER OUTCOMES:
Adverse events | up to one hour
  Any suspected or confirmed adverse events during and after recording of FiO2

CONTACTS AND LOCATIONS:
Locations (1):
- Phu San Hanoi Hospital, Hanoi, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the current study will be available from the principal investigator on reasonable request after publication of results.

REFERENCES:
- See also: WHO guidelines including respiratory care — https://www.who.int/publications/i/item/9789240058262